CLINICAL TRIAL: NCT00745134
Title: A Randomized Double Blinded Study of Curcumin With Pre-operative Capecitabine and Radiation Therapy Followed by Surgery for Rectal Cancer
Brief Title: Radiation Therapy and Capecitabine With or Without Curcumin Before Surgery in Treating Patients With Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped early because there was only one patient with pCR among the first 15 patients randomized to the curcumin arm.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2006-0644; NCI-2012-01676 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0644 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Rectal Mucinous Adenocarcinoma; Rectal Signet Ring Cell Adenocarcinoma; Recurrent Rectal Carcinoma; Stage IIA Rectal Cancer AJCC v7; Stage IIB Rectal Cancer AJCC v7; Stage IIC Rectal Cancer AJCC v7; Stage IIIA Rectal Cancer AJCC v7; Stage IIIB Rectal Cancer AJCC v7; Stage IIIC Rectal Cancer AJCC v7
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Curcumin; Radiotherapy; Radiation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (curcumin) (Experimental): Patients undergo radiation therapy 5 days a week for a total of 28 fractions. Patients also receive capecitabine PO BID on the days of radiation therapy and curcumin PO BID in weeks 1-11.5.
  Interventions: Drug: Capecitabine; Dietary Supplement: Curcumin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy
- Arm II (placebo) (Active Comparator): Patients undergo radiation therapy and receive capecitabine as in Arm I. Patients also receive placebo PO BID in weeks 1-11.5.
  Interventions: Drug: Capecitabine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Other: Placebo; Other: Quality-of-Life Assessment; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Dietary Supplement: Curcumin — Given PO
  Other Names: C.I. 75300; C.I. Natural Yellow 3; Diferuloylmethane; Turmeric Yellow
  Arms: Arm I (curcumin)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Optional correlative studies
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Irradiate; Irradiated; irradiation; Radiation; Radiotherapeutics; RADIOTHERAPY; RT; Therapy, Radiation

SUMMARY:
This randomized phase II trial studies how well radiation therapy and capecitabine with or without curcumin before surgery works in treating patients with rectal cancer. Drugs such as curcumin may make tumor cells more sensitive to radiation therapy. Drugs used in chemotherapy, such as capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy with radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. It is not yet known whether chemotherapy and radiation therapy is more effective with or without curcumin when given before surgery in patients with rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of a combination of capecitabine and radiation therapy with or without curcumin in locally advanced rectal cancer as assessed by pathological complete response rate.

SECONDARY OBJECTIVES:

I. To determine downstaging, local control, disease-free survival and overall survival rates.

II. To determine serum and rectal tumor tissue pharmacology of curcumin and its metabolites in the above patients and its correlation with clinical response.

III. To identify surrogate molecular markers for curcumin effects. IV. To correlate serum cytokine levels with quality of life in patients receiving this therapy.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients undergo radiation therapy 5 days a week for a total of 28 fractions. Patients also receive capecitabine orally (PO) twice daily (BID) on the days of radiation therapy and curcumin PO BID in weeks 1-11.5.

ARM II: Patients undergo radiation therapy and receive capecitabine as in Arm I. Patients also receive placebo PO BID in weeks 1-11.5.

After completion of study treatment, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have clinical stage T3,4 N0,1,2 or T2N1,2 adenocarcinoma of the rectum; patients will be clinically staged using endorectal ultrasound, pelvic computed tomography (CT) or magnetic resonance imaging (MRI), and physical examination
* Histology must be confirmed with review by the Department of Pathology at MD Anderson Cancer Center (MDACC)
* All patients must have no distant metastatic disease in the liver, peritoneum, lungs, or paraaortic lymph nodes
* Patients must have a performance status (Karnofsky scale) of 70% or greater
* Absolute neutrophil count (ANC) > 1200 cells/mm^3
* Platelets > 100,000/mm^3
* Total serum bilirubin < 2 mg/dl
* Blood urea nitrogen (BUN) < 30 mg/dl
* Creatinine < 1.5 mg/dl or creatinine clearance > 50cc/min (estimated as calculated with Cockcroft-Gault equation)
* Patients must have signed informed consent indicating that they are aware of the investigational nature of the study, and are aware that participation is voluntary; patients must also agree to refrain from use of additional herbal supplements during the course of the study
* Patients will agree to continue contraception for 30 days from the date of the last study drug administration; sexually active males must practice contraception during the study
* Postmenopausal woman must have been amenorrheic for at least 12 months to be considered of non-childbearing potential

Exclusion Criteria:

* Prior complete course up to 5 Gy of radiotherapy to the pelvis
* Pregnant or lactating woman; women of childbearing potential who have not undergone a hysterectomy with either a positive or no pregnancy test at baseline; women / men of childbearing potential not using a reliable and appropriate contraceptive method (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner)
* Treatment for other carcinomas within the last five years, except cured non-melanoma skin and treated in-situ cervical cancer
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or requiring IV antibiotics, cardiac disease New York Heart Association (NYHA) class III or IV, unstable angina pectoris, unstable cardiac arrhythmia or tachycardia (heart rate > 100 beats/minute), or psychiatric illness/ social situations that would limit compliance with the study requirements are excluded
* Other serious uncontrolled medical conditions that the investigator feels might compromise study participation
* Major surgery within 4 weeks of the start of study treatment
* Prior unanticipated severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil or capecitabine or curcumin
* Concurrent use of Coumadin other than low dose (1 mg) Coumadin used for line patency; patients on Coumadin must be changed to Lovenox at least 1 week prior to starting capecitabine
* Concurrent use of cimetidine, allopurinol, or aluminium hydroxide and magnesium hydroxide-containing antacids such as Maalox
* Sorivudine and brivudine use within 4 weeks of the start of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-08-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jillian R. Gunther, PHD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Gunther JR, Chadha AS, Guha S, Raju GS, Maru DM, Munsell MF, Jiang Y, Yang P, Felix E, Clemons M, Mathew GG, Singh PK, Skibber JM, Rodriguez-Bigas MA, Chang GJ, Eng C, Delclos ME, Crane CH, Das P, Krishnan S. A phase II randomized double blinded trial evaluating the efficacy of curcumin with pre-operative chemoradiation for rectal cancer. J Gastrointest Oncol. 2022 Dec;13(6):2938-2950. doi: 10.21037/jgo-22-259. PMID 36636059
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Curcumin): Participants received CRT [50.4 gray in 28 fractions; capecitabine (825 mg/m2 twice daily)] followed by surgery. Curcumin (4 grams orally, twice daily)
- Arm II (Placebo): Participants underwent radiation therapy and receive capecitabine as in Arm I. Patients also receive placebo PO BID in weeks 1-11.5.
Period: Overall Study
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Started | 15 | 7
Completed | 15 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Curcumin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 15 | 7 | 22
Age, Continuous [Median (Full Range); unit: years] | 69 [28 to 75] | 50 [45 to 64] | 60 [28 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 7 | 2 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 22
Clinical T (Tumor) Stage [Count of Participants; unit: Participants] — Refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues.
  Participants
    T2 | 3 | 1 | 4
    T3 | 11 | 6 | 17
    T4 | 1 | 0 | 1
Clinical N (Nodal) Stage [Count of Participants; unit: Participants] — Refers to the number and location of lymph nodes that contain cancer. The higher the number after the N, the more lymph nodes that contain cancer.
  Participants
    N0 | 3 | 3 | 6
    N1 | 11 | 4 | 15
    N2 | 1 | 0 | 1
Tumor Size [Median (Full Range); unit: cm] | 4 [2 to 8] | 5 [4 to 8] | 4.5 [2 to 8]
Distance from anal verge [Median (Full Range); unit: cm] | 3 [1 to 9] | 6.5 [2 to 10] | 4 [1 to 10]
Tumor circumference [Median (Full Range); unit: cm] | 50 [15 to 100] | 55 [40 to 75] | 50 [15 to 100]
Pretreatment Carcinoembryonic Antigen (CEA) [Median (Full Range); unit: ng/mL] | 1.3 [1 to 5.4] | 2.4 [1.0 to 8.1] | 1.6 [1.0 to 8.1]
Number of Participants with Tumor differentiation [Count of Participants; unit: Participants] — Well differentiated, low grade; Moderately differentiated, intermediate grade; Poorly differentiated, high grade
  Participants
    Well Differentiated | 0 | 0 | 0
    Moderately Differentiated | 15 | 7 | 22
    Poorly Differentiated | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pathologic Complete Response (pCR) Rate
Description: Compared the rate of pCR between treatment arms with Fisher's exact test.
Time Frame: At time of surgery
Measure: Count of Participants; unit: Participants
Groups:
- Arm I (Curcumin): Participants received chemoradiation therapy (CRT) [50.4 gray in 28 fractions; capecitabine (825 mg/m2 twice daily)] followed by surgery. Curcumin (4 grams orally, twice daily)
- Arm II (Placebo): Participants underwent radiation therapy and receive capecitabine as in Arm I. Participants received placebo PO BID in weeks 1-11.5.
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 7
Participants | 1 | 2

2. Secondary Outcome: Change in Curcumin Level in Tumor Tissue
Description: A logistic regression model with pCR as the dependent variable will be used to assess the association between pCR and NF-kB activity and treatment.
Time Frame: Baseline to 11.5 weeks
Population: Participants with analyzable tissue biopsies.
Measure: Median (Full Range); unit: ng/mg tissue
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 12 | 3
ng/mg tissue | 33.7 [0.1 to 4765.7] | 0.0 [0.0 to 0.0]

3. Secondary Outcome: Change in Curcumin Level in Serum
Description: Plasma levels were assessed pre and post curcumin/placebo administration. During week 2 (after at least 5 fractions of radiation therapy) of chemoradiation therapy:
  1. Optional endoscopic biopsy
  2. Optional blood collection for pharmacology (1 hour before and 1 hour after intake of curcumin or placebo)
Time Frame: assessed 1 hr pre/post curcumin administration on one of the days during week 2 of radiation therapy (fractions 6-10)
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm I (Curcumin)
Number analyzed (Participants) | 15
ng/mL
  Serum curcumin concentrations before curcumin/placebo administration. | 3.04 [1.24 to 18.88]
  Serum curcumin concentrations after curcumin/placebo administration. | 3.32 [0.84 to 5.36]
Statistical Analysis 1: Comparison: Arm I (Curcumin); Test type: Other; p = 0.33, ANOVA

4. Secondary Outcome: Tumor Regression Grade
Description: tumor regression grade (1= pCR, 2= near pCR, 3= partial response, 4= no response, 5=progression).
Time Frame: Baseline to 11.5 weeks
Population: One patient who did not undergo surgical resection was removed from analyses related to pathologic response outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 6
Participants
  Grade 1 | 1 | 2
  Grade 2 | 2 | 1
  Grade 3 | 4 | 1
  Grade 4 | 8 | 2
  Grade 5 | 0 | 0

5. Secondary Outcome: Overall Survival (OS)
Description: OS was calculated from start of CRT to date of death, censored at last follow-up. Estimated with the Kaplan-Meier method.
Time Frame: 5 years
Population: One patient who did not undergo surgical resection was removed from analyses related to pathologic response outcomes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 6
percentage of participants | 85.7 [69.2 to 100] | 85.7 [63.3 to 100]

6. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was calculated from start of CRT to date of disease progression or death, censored at last endoscopy/imaging evaluation.
Time Frame: 5 years
Population: One patient who did not undergo surgical resection was removed from analyses related to pathologic response outcomes.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 6
percentage of participants | 66.7 [46.6 to 95.3] | 71.4 [44.7 to 100]

7. Secondary Outcome: Number of Participants With Tumor Downstaging
Description: Tumor downstaging (DS) is defined as a decrease in the T stage of the primary tumor by at least 1.
Time Frame: Baseline to 11.5 weeks
Population: One patient who did not undergo surgical resection was removed from analyses related to pathologic response outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
Number analyzed (Participants) | 15 | 6
Participants | 7 | 4

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Arm I (Curcumin) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 6/15 | 2/7
Serious Adverse Events (participants affected / at risk) | 1/15 | 0/7
Other Adverse Events (participants affected / at risk) | 15/15 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Curcumin) (N=15) | Arm II (Placebo) (N=7)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) — due to radiation
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Curcumin) (N=15) | Arm II (Placebo) (N=7)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (9) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 12 (13) | 3 (3)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 5 (6) | 0 (0)
Elevated liver function tests (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 13 (13) | 6 (6)
Hand foot syndrome (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 4 (4)
Neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 9 (10) | 5 (7)
Radiation dermatitis (Injury, poisoning and procedural complications) | 12 (14) | 4 (6)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT00745134/Prot_SAP_000.pdf